CLINICAL TRIAL: NCT00243594
Title: Active Immunization of Patients With Stage III and IV Melanoma in Whom a Regional Lymph Node Dissection is Planned, With Peptide-Pulsed Dendritic Cells: Evaluation of in Vivo Immune and Clinical Response and Migration
Brief Title: Dendritic Cell Vaccination in Melanoma Patients Scheduled for Regional Lymph Node Dissection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: C.J.A. Punt, MD, PhD, Radboud University Nijmegen Medical Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-3126; 2004-3126; KUN99-1950
Record Dates: First submitted 2005-10-21; First posted 2005-10-24 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2009-02

CONDITIONS: Melanoma Stage III or IV
Keywords: Dendritic cells; Immunotherapy; Vaccination; Melanoma; Peptides; MRI; Scintigraphy; Immune response
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Peptide-pulsed dendritic cells — peptide-pulsed dendritic cells

SUMMARY:
Dendritic cells (DCs) are the professional antigen-presenting cells of the immune system. As such they are currently used in clinical vaccination protocols in cancer patients, and both immunological and clinical responses have been observed. For these therapies accurate delivery to target organs is essential. Correct delivery and subsequent migration of vaccinated DCs to regional lymph nodes is of paramount importance for effective stimulation of the immune system. Currently it is not known what the best route of administration is for DC vaccines.

Using magnetically labeled DCs, we investigate the potential of MRI cell tracking to monitor DC therapy. This is investigated in stage III/IV melanoma patients in whom a regional lymph node dissection is scheduled. Autologous monocyte-derived DCs are labeled with the clinically approved superparamagnetic iron oxide (SPIO) formulation Endorem and 111In-oxine and injected either in the skin or directly in lymph nodes under ultrasound guidance. Two days after vaccination patients are monitored with scintigraphy and MR imaging. Lymph nodes are then resected. Subsequently patients receive 3 more vaccination with DCs. During and after therapy immune responses against the used melanoma peptides are monitored.

ELIGIBILITY:
Inclusion criteria:

Histologically documented evidence of melanoma

Stage III-IV melanoma according to the 2001 AJCC criteria

Radical lymph node dissection planned, either with curative (stage III) or palliative (stage IV) intent

Melanoma expressing gp100 (compulsory) and tyrosinase (non-compulsory)

HLA-A2.1 phenotype according to lymphocyte HLA typing

ECOG performance status 0-1, life expectancy > 3 months

Age 18-75 years

Interval since last prior chemotherapy, immunotherapy or radiotherapy at least 4 weeks, no residual toxicity of prior treatment.

WBC > 3.0 x 109/l, lymphocytes > 0.8 x 109/l, platelets > 100 x 109/l, serum creatinine < 150 μmol/l, serum bilirubin < 25 μmol/l

Written informed consent

Expected adequacy of follow-up

Exclusion criteria:

No clinical signs of CNS metastases, in patients with a clinical suspicion of other metastases diagnostic tests should be performed to exclude this.

No concomitant use of corticosteroids or other immunosuppressive agents

No history of second malignancy within the last 5 years. Adequately treated basal carcinoma of skin or carcinoma in situ of cervix is acceptable within this period

No serious concomitant disease, no active infections. No autoimmune disease or organ allografts, no clinical suspicion of HIV or Hepatitis B

No contra-indications for MRI-scanning: claustrophobia, pacemaker or pacemaker threads, cerebral clips or artificial heartvalves, internal hearing prosthesis No known allergy to shell fish (contains KLH)

No pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 1999-09; Primary Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Immune response | during the first 10 years
Migration efficacy | during the first 1-2 years

SECONDARY OUTCOMES:
Clinical response | during the first 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Prof. C.J.A. Punt, MD, PhD, Principal Investigator — Radboud University Medical Center; Prof. C.G. Figdor, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, PO Box 9101, Netherlands

REFERENCES:
- [Background] de Vries IJ, Bernsen MR, Lesterhuis WJ, Scharenborg NM, Strijk SP, Gerritsen MJ, Ruiter DJ, Figdor CG, Punt CJ, Adema GJ. Immunomonitoring tumor-specific T cells in delayed-type hypersensitivity skin biopsies after dendritic cell vaccination correlates with clinical outcome. J Clin Oncol. 2005 Aug 20;23(24):5779-87. doi: 10.1200/JCO.2005.06.478. PMID 16110035
- [Background] Lesterhuis WJ, de Vries IJ, Adema GJ, Punt CJ. Dendritic cell-based vaccines in cancer immunotherapy: an update on clinical and immunological results. Ann Oncol. 2004;15 Suppl 4:iv145-51. doi: 10.1093/annonc/mdh919. No abstract available. PMID 15477299
- [Background] Figdor CG, de Vries IJ, Lesterhuis WJ, Melief CJ. Dendritic cell immunotherapy: mapping the way. Nat Med. 2004 May;10(5):475-80. doi: 10.1038/nm1039. PMID 15122249
- [Background] de Vries IJ, Lesterhuis WJ, Scharenborg NM, Engelen LP, Ruiter DJ, Gerritsen MJ, Croockewit S, Britten CM, Torensma R, Adema GJ, Figdor CG, Punt CJ. Maturation of dendritic cells is a prerequisite for inducing immune responses in advanced melanoma patients. Clin Cancer Res. 2003 Nov 1;9(14):5091-100. PMID 14613986
- [Background] De Vries IJ, Krooshoop DJ, Scharenborg NM, Lesterhuis WJ, Diepstra JH, Van Muijen GN, Strijk SP, Ruers TJ, Boerman OC, Oyen WJ, Adema GJ, Punt CJ, Figdor CG. Effective migration of antigen-pulsed dendritic cells to lymph nodes in melanoma patients is determined by their maturation state. Cancer Res. 2003 Jan 1;63(1):12-7. PMID 12517769
- [Background] de Vries IJ, Eggert AA, Scharenborg NM, Vissers JL, Lesterhuis WJ, Boerman OC, Punt CJ, Adema GJ, Figdor CG. Phenotypical and functional characterization of clinical grade dendritic cells. J Immunother. 2002 Sep-Oct;25(5):429-38. doi: 10.1097/00002371-200209000-00007. PMID 12218781
- [Background] Adema GJ, de Vries IJ, Punt CJ, Figdor CG. Migration of dendritic cell based cancer vaccines: in vivo veritas? Curr Opin Immunol. 2005 Apr;17(2):170-4. doi: 10.1016/j.coi.2005.01.004. PMID 15766677
- [Background] de Vries IJ, Lesterhuis WJ, Barentsz JO, Verdijk P, van Krieken JH, Boerman OC, Oyen WJ, Bonenkamp JJ, Boezeman JB, Adema GJ, Bulte JW, Scheenen TW, Punt CJ, Heerschap A, Figdor CG. Magnetic resonance tracking of dendritic cells in melanoma patients for monitoring of cellular therapy. Nat Biotechnol. 2005 Nov;23(11):1407-13. doi: 10.1038/nbt1154. Epub 2005 Oct 30. PMID 16258544
- [Derived] Aarntzen EH, Srinivas M, Bonetto F, Cruz LJ, Verdijk P, Schreibelt G, van de Rakt M, Lesterhuis WJ, van Riel M, Punt CJ, Adema GJ, Heerschap A, Figdor CG, Oyen WJ, de Vries IJ. Targeting of 111In-labeled dendritic cell human vaccines improved by reducing number of cells. Clin Cancer Res. 2013 Mar 15;19(6):1525-33. doi: 10.1158/1078-0432.CCR-12-1879. Epub 2013 Feb 4. PMID 23382117
- See also: Home page of the Radboud University Nijmegen Medical Centre — http://www.umcn.nl
- See also: Website of the department of Tumor Immunology of the Nijmegen Centre for Molecular Life Sciences of the Radboud University Nijmegen Medical Centre — http://www.ncmls.nl/